CLINICAL TRIAL: NCT01798355
Title: Children and Adolescents With Dental Anxiety - Randomized Controlled Study of Cognitive Behavioral Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Eastmaninstitutet (Other)
Responsible Party: Principal Investigator, Shervin Shahnavaz, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KIPED20130218
Record Dates: First submitted 2013-02-20; First posted 2013-02-25 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Dental Anxiety
Keywords: Dental Fear; Dental Phobia; Cognitive Behavior Therapy; Specific Phobia; Children and Adolescents anxiety; Self Efficacy
MeSH Terms: conditions — Phobia, Specific | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Treatment as usual (Active Comparator)
  Interventions: Behavioral: Treatment As Usual

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The treatment group is offered cognitive behavior therapy(CBT) by psychologists/psychotherapists. CBT is offered according to a treatment manual and consists of 10- sessions during 12-15 weeks.
  Arms: Cognitive Behavioral Therapy
Behavioral: Treatment As Usual — Treatment as usual consist of strategies such as habituation, tell-show-do, premedication with midazolam, nitrous oxide sedation and general anesthesia. All offered by dentists and dental hygienist and/or dental assistants.
  Arms: Treatment as usual

SUMMARY:
The purpose of this study is to determine whether cognitive behaviour therapy is effective in the treatment of children and adolescents with dental anxiety. Our hypothesis is that children and adolescents who have been offered CBT shows significant better performance on outcome measures compared with patients in control group who have received treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* The patient and parents agree to participate in the research project
* A primary diagnosis of specific phobia (dental anxiety or needle phobia) can be established according to the Diagnostic and Statistical Manual of Mental Disorders, 4th. Edition.

Exclusion Criteria:

* The diagnostic interview shows that other psychiatric or developmentally related diagnoses should be consider as the primary diagnosis
* The patient undergoing psychiatric examination and/or psychotherapy
* The patient has no dental treatment needs or the dental treatment needs are of an emergency nature.

Ages: 7 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Changes in dental anxiety | 3 months and 12 months from baseline
  Both child and parental versions of Children's Fear Survey Schedule - Dental Subscale will be administered.

SECONDARY OUTCOMES:
Changes in Behavioral Avoidance | 3 months and 12 months from baseline
  Behavioral Avoidance Test consists of 18 dental situations. The patient is exposed to a situation at a time. Patients receive 1 point for every step he / she manage. The test is stopped when the patient does not want to go further.

OTHER OUTCOMES:
General psychopathology | 3 months, 12 months from baseline
  Changes in general psychopathology is assessed by Developmental and Well-Being Assessment Questionnaire
Changes in Self efficacy | 3 months and 12 months from baseline
  Self Efficacy is assessed by the Self Efficacy Questionnaire for Specific Phobias

CONTACTS AND LOCATIONS:
Overall Officials: Göran Dahllöf, PhD, Study Director — Department of Dental Medicine, Karolinska Institutet; Shervin Shahnaavz, PhD, Principal Investigator — Department of Dental Medicine, Karolinska Institutet
Locations (1):
- Pediatric Dentistry, Department of Dental Medicine, Karolinska Institutet, Stockholm, Huddinge, Sweden

REFERENCES:
- [Background] Shahnavaz S, Hedman E, Grindefjord M, Reuterskiold L, Dahllof G. Cognitive Behavioral Therapy for Children with Dental Anxiety: A Randomized Controlled Trial. JDR Clin Trans Res. 2016 Oct;1(3):234-243. doi: 10.1177/2380084416661473. Epub 2016 Aug 15. PMID 29417092
- [Background] Shahnavaz S, Hedman-Lagerlof E, Hasselblad T, Reuterskiold L, Kaldo V, Dahllof G. Internet-Based Cognitive Behavioral Therapy for Children and Adolescents With Dental Anxiety: Open Trial. J Med Internet Res. 2018 Jan 22;20(1):e12. doi: 10.2196/jmir.7803. PMID 29358158
- [Background] Shahnavaz S, Rutley S, Larsson K, Dahllof G. Children and parents' experiences of cognitive behavioral therapy for dental anxiety--a qualitative study. Int J Paediatr Dent. 2015 Sep;25(5):317-26. doi: 10.1111/ipd.12181. Epub 2015 Jul 4. PMID 26147012
- See also: Registration website for our study of Internet-based CBT for pediatric dentala anxiety study — http://ki.se/dentmed/kbt